CLINICAL TRIAL: NCT06997406
Title: Explore the Benefit of 'Inner Ear Support' Oral Capsule in Patients With Sudden Sensorineural Hearing Loss - A Randomized, Open-label, Single-center Study
Brief Title: 'Inner Ear Support' Oral Capsule in Patients With Sudden Sensorineural Hearing Loss
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Far East Bio-Tec Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE-NTUH-FB1603
Record Dates: First submitted 2025-05-13; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Sudden Sensorineural Hearing Loss (SSNHL); Tinnitus
Keywords: Sudden Sensorineural Hearing Loss; SSNHL; C-phycocyanin; Tinnitus; Hearing Recovery; Inner Ear Support; Arthrospira; herbal medicine
MeSH Terms: conditions — Hearing Loss, Sudden; Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stand treatment (No Intervention): Based on clinical symptoms and the patient's physical condition, standard treatment will be provided, including the use of steroids (oral and/or intratympanic injection) and hyperbaric oxygen therapy.
- stand treatment +Inner ear support (Experimental): Based on clinical symptoms and the patient's physical condition, standard treatment will be provided, including the use of steroids (oral and/or intratympanic injection) and hyperbaric oxygen therapy. In addition, subjects will take 'Inner ear support' oral capsules in the morning and evening (600 mg per dose, 1200 mg per day).
  Interventions: Dietary Supplement: Inner ear support

INTERVENTIONS:
Dietary Supplement: Inner ear support — FB-1603 (150 mg): A cold water extract of Arthrospira maxima (a species of blue-green algae), rich in the antioxidant pigment C-phycocyanin (C-PC).
  GABA (126 mg): A natural calming neurotransmitter that can help reduce nerve-related overactivity.
  γ-Oryzanol (12 mg): A component from rice bran oil, known for its antioxidant properties.
  Sesamin (12 mg): A compound from sesame seeds, with potential neuroprotective and anti-inflammatory benefits.
  Arms: stand treatment +Inner ear support

SUMMARY:
Sudden sensorineural hearing loss (SSNHL) is a medical condition where people experience rapid hearing loss, usually in one ear, over a short period of time (typically within 72 hours). It can affect people of any age, though it is more common among adults aged 40 to 60. In many cases, the exact cause remains unknown, but possible reasons include viral infections, immune-related problems, and reduced blood circulation to the inner ear. Along with hearing loss, many patients may also experience tinnitus (ringing in the ears) or dizziness.

The standard treatment for SSNHL often involves steroids, sometimes combined with hyperbaric oxygen therapy. However, the effectiveness of these treatments varies, and many patients do not fully recover their hearing. This study aims to explore whether an additional supplement-'Inner ear support' oral capsule-can improve hearing outcomes and relieve associated symptoms in patients with SSNHL.

The study will involve 80 participants who are randomly assigned to two groups. Both groups will receive standard treatment (including steroids and possibly hyperbaric oxygen therapy), but only the test group will take the 'Inner ear support' capsule twice daily for 28 days. Participants will be followed and evaluated over a period of 196 days through hearing tests and symptom questionnaires.

'Inner ear support' is a commercially available nutritional supplement that includes FB-1603 (an extract from Arthrospira maxima), GABA, gamma-oryzanol, and sesamin. Previous research has shown that FB-1603 and its active component, C-phycocyanin, have anti-inflammatory, antioxidant, and nerve-protective effects. Animal studies suggest it may help reduce tinnitus and prevent hearing deterioration.

This clinical trial is designed to evaluate whether 'Inner ear support' can enhance hearing recovery, improve tinnitus and dizziness symptoms, and be safely used as an additional treatment in patients with sudden hearing loss. All participants will be monitored for any potential side effects during the study period.

The ultimate goal of this study is to determine whether' Inner ear support' could become a helpful addition to current treatment methods for SSNHL, improving patient outcomes and quality of life.

DETAILED DESCRIPTION:
Sudden sensorineural hearing loss (SSNHL) is an otologic emergency characterized by rapid onset of hearing loss, typically unilateral, occurring over less than 72 hours. The annual incidence is estimated to range from 5 to 30 per 100,000 individuals, with the highest prevalence among adults aged 40-60. The etiology of SSNHL remains idiopathic in most cases, though proposed mechanisms include viral infections, autoimmune responses, vascular compromise, or membrane rupture in the inner ear. In addition to hearing loss, patients commonly report tinnitus, ear fullness, and vertigo, which may significantly affect quality of life.

Standard treatment modalities for SSNHL include systemic corticosteroids and, in moderate to severe cases, hyperbaric oxygen therapy. However, current literature indicates that only approximately 60% of patients achieve significant improvement, leaving a substantial proportion with residual deficits. There remains an unmet need for adjunctive therapies that are both effective and safe.

The investigational product in this study is 'Inner ear support' oral capsule, a commercially available dietary supplement composed of FB-1603 (a cold water extract of Arthrospira maxima), gamma-aminobutyric acid (GABA), gamma-oryzanol, and sesamin. Among these, FB-1603 contains biologically active compounds such as C-phycocyanin, a pigment-protein complex that has demonstrated antioxidant, anti-inflammatory, and neuroprotective properties in preclinical studies.

In vitro studies show that FB-1603 significantly reduces LPS-induced cytotoxicity and suppresses the expression of pro-inflammatory markers such as iNOS, COX-2, TNF-α, and IL-6 in BV-2 microglial cells. Animal studies using salicylate-induced tinnitus models in mice have demonstrated that dietary supplementation with FB-1603 or C-phycocyanin attenuates the expression of auditory-related inflammatory genes (e.g., TNF-α, IL-1β, COX-2, NR2B) in the cochlea and inferior colliculus.

Additional preclinical evidence suggests that FB-1603 modulates the expression of ion transporters such as KCC2 and NKCC1, potentially restoring auditory neural excitability. In senescence-accelerated mouse models, FB-1603 was found to enhance antioxidant enzyme expression (SOD, catalase, GPx), suggesting a protective role against age-related hearing decline. These findings form the basis for evaluating FB-1603 as a candidate therapeutic agent for sensorineural hearing dysfunction.

This randomized, open-label, single-center clinical trial aims to evaluate the efficacy and safety of 'Inner ear support' oral capsule in patients with SSNHL. A total of 80 patients will be enrolled and randomly assigned to two groups: both will receive standard treatment with systemic corticosteroids (with or without hyperbaric oxygen), but only the experimental group will receive 'Inner ear support' 600 mg daily (administered as two 300 mg capsules per day) for 28 days.

The primary endpoint is the change in pure tone audiometry (PTA) thresholds from baseline at Days 28, 84, and 168. Secondary endpoints include the incidence of adverse events, changes in clinical laboratory parameters (hematology, biochemistry, ECG), and patient-reported outcomes such as the Tinnitus Functional Index (TFI) and Dizziness Handicap Index (DHI).

All participants will undergo safety monitoring, and any adverse events will be recorded and evaluated. The study hypothesis is that 'Inner ear support', when added to standard treatment, will improve auditory recovery and reduce the severity of associated symptoms such as tinnitus and dizziness, without introducing significant safety risks.

This investigation will provide essential clinical data regarding the utility of a plant-derived, nutraceutical formulation as a novel adjunctive approach to managing SSNHL. If successful, 'Inner ear support' could offer a safe, accessible option to improve outcomes for patients affected by this disabling condition.

Study Design and Visit Schedule

This is a randomized, open-label, single-center clinical study. A total of 80 participants diagnosed with SSNHL will be randomly assigned in a 1:1 ratio to either the experimental group or the control group. Both groups will receive standard-of-care treatment including systemic corticosteroids, and, if clinically indicated, hyperbaric oxygen therapy. The experimental group will additionally receive 'Inner ear support' oral capsule at a dose of 300 mg twice daily for 28 days.

Participants will be evaluated at baseline (Day 0) and subsequently on Days 28, 84, and 168. Each visit will include:

* Pure tone audiometry (PTA)
* Laboratory tests (hematology, biochemistry)
* Electrocardiogram (ECG)
* Tinnitus Functional Index (TFI)
* Dizziness Handicap Index (DHI)
* Adverse event and safety assessments

Compliance and concomitant medication usage will also be recorded. Audiologic tests will follow standard frequencies (e.g., 0.5, 1, 2, and 4 kHz), and hearing threshold changes will be calculated as the mean difference compared to baseline.

Pharmacological Mechanism and Molecular Action of 'Inner ear support'

The primary active ingredient in 'Inner ear support' is FB-1603, a cold water extract of Arthrospira maxima, rich in the pigment C-phycocyanin (C-PC). C-PC exerts antioxidant and anti-inflammatory effects via several mechanisms:

* Suppression of oxidative stress: FB-1603 upregulates antioxidant enzymes such as superoxide dismutase (SOD), catalase, and glutathione peroxidase, reducing reactive oxygen species (ROS) in cochlear and brainstem tissues.
* Neuroprotection: C-PC inhibits pro-inflammatory cytokines (TNF-α, IL-6, IL-1β) and enzymes like iNOS and COX-2, preserving neural integrity under oxidative or inflammatory stress.
* Modulation of ion transport: FB-1603 downregulates aberrant expression of potassium-chloride co-transporter KCC2, implicated in auditory hypersensitivity and tinnitus, restoring synaptic excitability.

These actions are supported by in vivo studies in mouse models of salicylate-induced tinnitus and age-related hearing loss, where FB-1603 administration reduced auditory threshold shifts, inflammation-related gene expression, and tinnitus behavioral scores.

Statistical Analysis

This study will primarily employ:

* Paired and independent t-tests to assess changes in pure tone audiometry (PTA) between and within groups at multiple timepoints (Days 28, 84, 168).
* Chi-square tests for categorical data such as the proportion of patients with clinically significant improvement in hearing or symptom scores (TFI, DHI).
* All p-values will be two-sided, with a significance level set at α = 0.05.

Descriptive statistics (mean, standard deviation, range) will be presented for all quantitative outcomes. Safety analysis will summarize adverse events by type, severity, and relationship to the investigational product. Missing data will be handled using intention-to-treat principles; sensitivity analyses may be performed to evaluate robustness.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years
* Patients diagnosed with sudden sensorineural hearing loss as determined by the principal or sub-investigator
* Average hearing threshold in the affected ear ≥ 60 dB
* Initiation of treatment within two weeks of hearing loss onset

Exclusion Criteria:

* Patients with congenital or hereditary hearing loss
* Patients with fluctuating hearing loss
* Patients currently participating in other interventional treatments for sudden hearing loss
* Patients who have undergone surgery on the affected ear
* Patients with neurological or psychiatric disorders
* Patients with heart failure or ischemic heart disease
* Patients with immunodeficiency
* Patients with vestibular schwannoma (acoustic neuroma)
* Patients with other internal medical conditions deemed by the investigator to potentially interfere with the study conduct or outcomes
* Pregnant patients
* Patients with a known allergy to the investigational product
* Patients currently using acetylcysteine or products containing ginkgo biloba extract
* Patients with autoimmune diseases or currently receiving immunosuppressive therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in pure tone audiometry (PTA) | Baseline (Day 0), V2 (Day 28), V3 (Day 84), and V4 (Day 168)
  Changes in pure tone audiometry (PTA) results at V2 (Day 28), V3 (Day 84), and V4 (Day 168) compared to baseline.

SECONDARY OUTCOMES:
Change in AST (Aspartate Transaminase) level from baseline | Baseline (Day 0), V2 (Day 28), V3 (Day 84), and V4 (Day 168)
  Mean change in serum AST level (U/L) from baseline to V2 (Day 28), V3 (Day 84), and V4 (Day 168).
Change in ALT (Alanine Transaminase) level from baseline | Baseline (Day 0), V2 (Day 28), V3 (Day 84), and V4 (Day 168)
  Mean change in serum ALT level (U/L) from baseline to V2, V3, and V4.
Change in serum albumin level from baseline | Baseline (Day 0), V2 (Day 28), V3 (Day 84), and V4 (Day 168)
  Mean change in serum albumin concentration (g/dL) from baseline to V2, V3, and V4.
Change in alkaline phosphatase (Alk-P) level from baseline | Baseline (Day 0), V2 (Day 28), V3 (Day 84), and V4 (Day 168)
  Mean change in serum alkaline phosphatase level (U/L) from baseline to V2, V3, and V4.
Change in gamma-glutamyl transpeptidase (GGT) level from baseline | Baseline (Day 0), V2 (Day 28), V3 (Day 84), and V4 (Day 168)
  Mean change in serum GGT (gamma-GT) level (U/L) from baseline to V2, V3, and V4.
Change in total protein level from baseline | Baseline (Day 0), V2 (Day 28), V3 (Day 84), and V4 (Day 168)
  Mean change in serum total protein concentration (g/dL) from baseline to V2, V3, and V4.
Changes in Tinnitus Functional Index (TFI) | Baseline (Day 0), V2 (Day 28), V3 (Day 84), and V4 (Day 168)
  Changes in Tinnitus Functional Index (TFI) at V2 (Day 28), V3 (Day 84), and V4 (Day 168) compared to baseline.
  The Tinnitus Functional Index (TFI) scoring uses a scale from 0 to 10 for each question and total 25 questions. (Total scoring from 0 to 250)
  TFI Scoring:
  0-43: Minimal or no problem. 43-79: Small problem. 79-134: Moderate problem. 134-180: Big problem. 180-250: Very big problem.
Changes in Dizziness Handicap Index (DHI) | Baseline (Day 0), V2 (Day 28), V3 (Day 84), and V4 (Day 168)
  Changes in Dizziness Handicap Index (DHI) at V2 (Day 28), V3 (Day 84), and V4 (Day 168) compared to baseline.
  The DHI is a 25-item self-reported measure with three categories: functional, emotional, and physical. It is an efficient outcome measure. The subject rates their perceived disability due to their dizziness by answering each question with - yes, sometimes, or no. The measure is then scored with points for each answer: No = 0, Sometimes = 2, and Yes = 4 points, thus the greater the score, the greater the perceived disability out of a total of 100 points.
  Further classification of scoring includes:
  Mild Handicap: 16-34 Points Moderate Handicap: 36-52 Points Severe Handicap: 54+ Points

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Hsuan Lin, P.h.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan